CLINICAL TRIAL: NCT01218737
Title: Double-Masked, Randomized, Parallel Group Study for Evaluation of Non-Inferiority of 0.3%Gatifloxacin/1.0% Prednisolone Association Compared With Their Isolated Administration in the Prevention of Ocular Infection/Inflammation After LASIK Surgery
Brief Title: Non-Inferiority of Gatifloxacin/Prednisolone Association vs Isolated Administration in Prevention of Ocular Infection/Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG9890X-001
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2010-10

CONDITIONS: Ocular Infection and Inflammation
MeSH Terms: conditions — Eye Infections; Inflammation | interventions — Gatifloxacin; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Association (Experimental): 0.3% gatifloxacin and 1.0% prednisolone acetate association in eye drops plus placebo
  Interventions: Drug: 0.3% gatifloxacin and 1.0% prednisolone acetate association
- Isolated ingredients (Active Comparator): 0.3% gatifloxacin and 1.0% prednisolone acetate isolated eye drops formulations
  Interventions: Drug: isolated 0.3% gatifloxacin and 1.0% prednisolone acetate

INTERVENTIONS:
Drug: 0.3% gatifloxacin and 1.0% prednisolone acetate association — Each patient will receive two medication bottles (eye drops) in a blinded fashion: one with the association and another with placebo. The patient must instill 01 drop of each bottle in each operated eye, with a 5-minute interval between the instillations.
  This procedure should be performed 4 times a day (QID) during the wake hours, from Day 0 (surgery day) until Day 15.
  Other Names: Zypred
  Arms: Association
Drug: isolated 0.3% gatifloxacin and 1.0% prednisolone acetate — Each patient will receive two medication bottles (eye drops) in a blinded fashion: one with the 0.3% gatifloxacin eye drops and another with 1.0% prednisolone acetate eye drops. The patient must instill 01 drop of each bottle in each operated eye, with a 5-minute interval between the instillations.
  This procedure should be performed 4 times a day (QID) during the wake hours, from Day 0 (surgery day) until Day 15.
  Other Names: Zymar; Pred Fort
  Arms: Isolated ingredients

SUMMARY:
The purpose of the study is to evaluate the safety and tolerance of the 0.3% gatifloxacin and 1.0% prednisolone acetate association in eye drops in the prevention of infection and inflammation after refractive surgery (Lasik) and also demonstrate the non-inferiority of the efficacy of this association compared to the administration of 0.3% gatifloxacin and 1.0% prednisolone acetate as isolated eye drops formulations. The study treatment is randomized, double-masked, with 2 parallel arms. Each patient's participation lasts 29 days, with 15 days of study treatment administration after the ocular surgery is performed. Candidates for the study are patients with indication for ocular refractive surgery (Lasik) for correction of visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated to have an ocular refractive surgery performed (myopia, astigmatism, hypermetropy) by the Lasik method.
* Patient presents a normal eye fundus.
* Patient has intraocular pressure (IOP) ≤ 20 mmHg.

Exclusion Criteria:

* Surgery and/or previous ocular pathology (presence of scar/change in the cornea, glaucoma, retinopathies, etc.).
* Patient has diabetes or is immunodepressed.
* Any systemic infection during the study.
* Signs and/or symptoms of ocular inflammation/infection (bacterial, viral, fungal, caused by Chlamydia, by Mycobacterium, Acanthamoeba or of allergic etiology).
* Have used any systemic or topical antibiotics for ocular infection in the previous 14 days.
* Patient has known hypersensitivity to any of the components of the formulations used in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percentage of eyes with absence of signs/symptoms of ocular infection/inflammation after surgery. | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Federal University of Sao Paulo - Dept of Ophthalmology, São Paulo, São Paulo, Brazil